CLINICAL TRIAL: NCT07191860
Title: A Randomized, Controlled, Multi-Center, Prospective Trial of Paclitaxel-Coated Pulmonary Balloon for the Treatment of Benign Airway Stenosis (OXYGEN-RCT Trial)
Brief Title: Paclitaxel-Coated Pulmonary Balloon for the Treatment of Benign Central Airway Stenosis
Acronym: OXYGEN-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Airiver Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol Number: PR3050
Record Dates: First submitted 2025-08-11; First posted 2025-09-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Adult Subjects With Symptomatic Benign Airway Obstruction; Adult Benign Central Airway Stenosis; Adult Tracheobronchial Stenosis; Tracheal Stenosis; Central Airway Stenosis; Central Airway Obstruction
MeSH Terms: conditions — Tracheal Stenosis | interventions — Dilatation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- treatment with the Airiver Pulmonary DCB (Experimental): dilate benign stenoses of the airway tree.
  Interventions: Combination Product: The Airiver Pulmonary drug-coated balloon (DCB) dilation
- treatment of Commercial airway dilation balloon (Active Comparator): dilate benign stenoses of the airway tree.
  Interventions: Device: Commercial airway balloon dilation

INTERVENTIONS:
Combination Product: The Airiver Pulmonary drug-coated balloon (DCB) dilation — drug coated balloon dilation
  Arms: treatment with the Airiver Pulmonary DCB
Device: Commercial airway balloon dilation — uncoated airway balloon dilation
  Arms: treatment of Commercial airway dilation balloon

SUMMARY:
The OXYGEN-RCT trial is a randomized, controlled, double blinded, prospective, multi-center trial to demonstrate the safety and efficacy in adult benign central airway stenosis. Participates will be in a 1:1 allocation to treatment with the Airiver Pulmonary DCB or standard of care laryngoscopic/bronchoscopic balloon dilation, respectively.

DETAILED DESCRIPTION:
Subjects will complete follow-up post-treatment at 30 days, 3 months, 6 months, 12 months, and every 6 months after through the primary endpoint, with a minimum of 2 years at study end.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 22 years.
2. Symptomatic de-novo or restenotic benign central airway stenosis in the subglottis, trachea, or mainstem bronchi with at least 50% narrowing, as determined by CT or bronchoscopy.
3. In the opinion of the investigator, subject can undergo laryngoscopy/bronchoscopy under general anesthesia and has a central airway stenosis amenable to balloon dilation.
4. For idiopathic subglottic stenoses, either de-novo or a dilation interval equal to or less than 18 months.
5. Target benign stenosis etiologies including:

   1. Post-intubation stenosis,
   2. Idiopathic subglottic stenosis,
   3. Post-transplantation stenosis,
   4. Non-malignant trachea-bronchial stenosis
6. Willing and able to complete protocol required follow-up visits.
7. Willing and able to provide written informed consent.

Exclusion Criteria:1. Two or more clinically significant (e.g. non-traversable) stenoses with total length >5cm or unable to be treated with a single balloon 2. Female subjects who are pregnant or breastfeeding or plan to become pregnant in next 12 months 3. Subject currently has a stent at target stenosis location or has had a stent at the target location within the past 90 days.

4. Subject has existing tracheostomy or had a tracheostomy within past 90 days 5. Contraindication to laryngoscopy/bronchoscopy, anesthesia, or deep sedation 6. Planned tracheal resection in the next 90 days. 7. Dynamic etiology of benign stenosis such as excessive dynamic airway collapse, tracheobronchomalacia, or stenosis due to external compression, or past tracheostomy which requires stent placement or surgical referral 8. Inclusion of vocal cord in target stenosis 9. Known medically significant unresolved lower respiratory tract infection, such as pneumonia, fungus, tuberculosis, etc.unrelated to stenosis 10. Target stenosis is beyond the mainstem bronchi 11. Signs or suspicion of a malignant airway obstruction NOTE: If obstruction is suspicious for malignancy based on clinical or laryngoscopic/bronchoscopic presentation, malignancy must be excluded by biopsy prior to randomization 12. Severe coagulation disorders or current use of anticoagulant or antiplatelet medication that cannot be safely managed per recommended guidelines prior to the index procedure 13. Chronic steroid use exceeding more than 10 mg per day for any medical condition including immunosuppression post-lung transplant or autoimmune associated airway suppression.

14. Received local steroid or chemotherapeutic treatments into target stenosis in the last 12 weeks or planned treatment during index or staged study procedure.

15. Planned serial intralesional steroid injections (SILSIs) post index procedure.

16. Stenosis not amenable to laryngoscopic/bronchoscopic dilation in the opinion of the investigator 17. Acute condition that requires emergent procedure prior to screening assessment 18. Concurrent medical condition that would affect the investigator's ability to evaluate the patient's condition or could compromise patient safety, such as recent myocardial infarction, severe pulmonary disease, bleeding diathesis, large thoracic aneurysm, pharyngeal or cervical deformity, ongoing infection, etc 19. Subject has known fistula between tracheobronchial tree and esophagus, mediastinum to pleural space.

20. Subject has vasculitis that is not well controlled in the opinion of the investigator.

21. Diagnosed with a disease requiring chemotherapy (e.g. cancer). 22. Allergy to paclitaxel or structurally related compounds 23. Target stenosis is within a transplanted lung or transplant anastomosis, or a tracheal resection anastomosis, which has been transplanted or resected within the last 60 days.

24. Target stenosis is related to radiation therapy 25. Subject has a life expectancy of less than 2 years. 26. Current participation in another pre-market drug or medical device clinical study that has not reached its primary endpoint.

-

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety: defined as Incidence of device- and/or procedure-related Major Adverse Events(MAEs) | 30 days post index procedure
  including:
  * Pneumothorax
  * Pneumomediastinum
  * Tracheal or bronchial laceration requiring intervention
  * Airway perforation or rupture
  * Required tracheostomy
  * Bleeding from treatment site consistent with massive hemoptysis defined as > 100mL of blood expectorated in 24 hours or requiring transfusion
  * Mediastinitis requiring the need for IV antibiotics and / or hospitalization
  * Respiratory distress or asphyxia requiring intubation or reintervention
  * Death
Primary Efficacy: freedom from clinically indicated target lesion re-intervention over time | Through the study completion, an average of 1 year
  defined as a therapeutic reintervention/dilation that occurs due to either a recurrence of patient symptoms due to the stenosis and/or a recurrence seen through imaging of the stenosis (≥ 50%) or is an emergent condition related to the stenosis and treatment is required.

SECONDARY OUTCOMES:
Time to first reintervention, defined as duration in days between the index/staged procedure and the first, subsequent procedure for treatment of the target stenosis. | From Day 1 until the date of first documented reintervention, assessed through the study completion, an average of 1 year.
  Hypothesis-test
Percent change in airway lumen area at 6 months by CT | Baseline, 6 months
  Hypothesis-test. The percent change expressed as the airway lumen volume within the treated segment at 6 months (Area 6mo), compared to the personal baseline airway lumen volume (AreaBL) on CT scan. Percent change in airway luminal area = (Area6mo - AreaBL) / AreaBL ×100%
Change in Peak Expiratory Flow (PEF) from 30 days to 6 months | 1 month, 6 months
  Hypothesis-test. PEF in L/min
Index procedure success, defined as the ability to deliver study device to the targeted stenosis, inflate, deflate, and remove and with a < 25% residual stenosis. | On index procedure day 0
  Non-hypothesis test. NO device malfunction issues. Use visual estimation under bronchoscopy at the end of index procedure, compare post-treated airway diameter (TD, mm) versus airway native diameter (ND, mm), residual stenosis = (ND- TD)/NDx100%
Change in airway lumen volume by CT at follow-up visit | Baseline, 30 days, 6 months, 12 months, then every 6 months until the date of the study complete (assessed up to 2 years)
  Non-hypothesis test. Change in lumen volume in percentage (%). The percent change expressed as the airway lumen volume within the treated segment at follow-up (AreaFU) compared to the personal baseline airway lumen volume (AreaBL) on CT scan. Percent change in airway luminal area = (AreaFU - AreaBL) / AreaBL ×100%
Freedom from reintervention, defined as any reintervention on the target stenosis, whether clinically indicated or not | 30 days, 3 months, 6 months, 12 months, then every 6 months until the date of study complete (assessed up to 2 years)
  Non-hypothesis test
Annualized rate, of reinterventions | Assessed annually through the date of the study complete, an average of 1 year.
  Non-hypothesis test
Secondary patency, defined as freedom from reintervention after a first reintervention, at each follow-up | From the date of the first reintervention to the next follow-up visit through the study completion, an average of 1 year.
  Non-hypothesis test
Change in forced expiratory volume in 1 second (FEV1) at follow-up visit | Baseline, 30 days, 3 months, 6 months, 12 months, then every 6 months until the date for the study complete (assessed up to 2 years)
  Non-hypothesis test. FEV1 in liters
Change in forced vital capacity (FVC) at follow-up visit | Baseline, 30 day, 3 months, 6 months, 12 months, then every 6 months until the date of the study complete (assessed up to 2 years)
  Non-hypnoses test. FVC in liters
Changes in the ratio of FVE1 and FVC at follow-up visit | Baseline, 30 days, 3 months, 6 months, 12 months, then every 6 months until the date of the study complete (assessed up to 2 years)
  Non-hypnoses test. The Ratio =(FVE1/FVC) x100%
Change in peak expiratory flow (PEF) | Baseline, 3 months, 12 months, then every 6 months until the date of the study complete (assessed up to 2 years).
  Non-hypnoses test. PEF in liters per minute (L/min)
Change in expiratory disproportion index (EDI) | Baseline, 30 days, 3 months, 6 months, 12 months, then every 6month until the date of the study complete (assessed up to 2 years)
  Non-hypnoses test. EDI= (FEV1/PEF) x100%
Rate of cannulation, stent, or open surgery due to target lesion stenosis | 30 days, 3 months, 6 months, 12 months, then every 6 months until the date of study complete (assessed up to 2 years)
  Non-hypothesis test
Change in modified Medical Research Council (mMRC) Dyspnea Scale | Baseline, 30 days, 3 months, 6 months, 12 months, then every 6 months until the date of study completion (assessed up to 2 years)
  Non-hypothesis test. mMRC is a self-assessment tool and rated on a scale from 0 to 4, where a higher score means a worse outcome.
Change in Chronic Obstructive Pulmonary Disease (COPD) Questionnaire | Baseline, 30 days, 3 months, 6 months, 12 months, then every 6 months until the date of study completion (assessed up to 2 years)
  Non-hypnoses test. The questionnaire is rated on 0-6 scale, a higher score indicating a worse health status.
Change in 12-Item Short Form (SF-12) Survey Global Quality of Life Score | Baseline, 30 days, 3 months, 6 months, 12 months, then every 6 months until the date of the study completion (assessed up to 2 years)
  Non-hypnosis test. SF-12 is a self-reported outcome and rated on a 0-5 scale, where a higher score indicates better health.
Change in Voice Handicap Index (VHI-10) questionnaire | Baseline, 30 days, 3 months, 6 months, 12 months, then every 6 months until the study completion (assessed up to 2 years)
  Non-hypnosis test. VHI-10 is a self-administered questionnaire and scored from 0 to 4, where a higher score indicates a greater voice -related handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hillel, MD, Principal Investigator — Johns Hopkins University; Ryan M Kern, MD, Principal Investigator — Mayo Clinic